CLINICAL TRIAL: NCT05843370
Title: Modification of Ambient Air Pollution Exposure and Cardiopulmonary Outcomes by Socioeconomic Status and Nutrition
Acronym: SENSE
Status: Enrolling by invitation | Type: Observational
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Haiyan Tong, Principal Investigator, Environmental Protection Agency (EPA)
Other Study IDs: 23-0428
Record Dates: First submitted 2023-03-24; First posted 2023-05-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Air Pollution; Pollution; Exposure; Nutrition, Healthy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High SVI: Participants reside in neighborhood zip code clusters that rank at the top of the social vulnerability index (most vulnerable)
- Low SVI: Participants reside in neighborhood zip code clusters that rank at the bottom of the social vulnerability index (least vulnerable)

SUMMARY:
The goal of this observational study is to compare the effects of air pollution exposure and nutrition between neighborhoods with high and low social vulnerability scores. The main questions this study aims to answer are:

* Does living in a neighborhood with high or low vulnerability influence the response of the heart, lungs, and immune system to air pollution.
* Does nutritional status alter the association between air pollution exposure and changes in the heart, lungs, and immune system.

Participants (age 25-70 years) that live in neighborhoods ranked high or low on the Social Vulnerability Index (SVI) will take part in 3 visits. Each visit involves the following:

* Measurements of heart activity, lung function, and blood to measure changes that may be caused by air pollution.
* Questionnaires about the types of food eaten and activities that may modify exposure to air pollution.
* Estimation of air pollution exposure using a study iPhone. Participants will carry a study iPhone with them for 24 hours at each visit. The study iPhone runs an application (app) that estimates the amount of air pollution each participant is exposed to.
* Wearing silicone wristbands for a week before each study visit. Silicone wristbands absorb air pollutants and are later measured see the types and amounts of chemicals participants are exposed to.

DETAILED DESCRIPTION:
Acute and chronic exposure to air pollution are well-established risk factors for all-cause mortality, mainly driven by cardiovascular and respiratory disease. The health effects of air pollution exposure have been shown to be mediated by a range of community level and personal factors, including the presence of preexisting medical conditions, age, and socioeconomic status (SES). Individuals who reside in lower SES communities are more likely to experience increased air pollution. The effects of air pollution among those residing in less advantaged communities may be further compounded by reduced access to health care and access to nutrition. Research conducted in our facility and others has established that increased levels of micronutrients can improve subclinical indices of cardiopulmonary disease after acute and chronic air pollution. Omega-3 polyunsaturated fatty acids (PUFAs) have been demonstrated to reduce the markers of cardiopulmonary dysfunction, including heart rate variability, cholesterol, and vascular injury markers after air pollution exposure. However, levels of PUFAs, as well as other potentially protective vitamins, have been demonstrated to be significantly reduced among individuals with lower income and lower educational attainment. This may be in part due to reduced access to healthy food options, as lower income and lower educational attainment have been shown to influence access to grocery stores and nutritious foods.

Given the interplay between nutrition, air pollution exposure, SES, and cardiopulmonary disease, the investigators propose the following study to investigate how socioeconomic status can modify ambient air pollution exposure and subclinical indices of cardiovascular and pulmonary disease and inflammation, and if nutritional status can further modify this relationship. Healthy 25-70-year- old male and female subjects will be recruited from communities that are representative of high and low social vulnerability index, a composite measure of urbanicity, educational attainment, owner-occupied housing, poverty, unemployment, non-managerial occupations, single parent households, houses built since 2000, vehicle ownership, and percentage of people who pay <30% of their income on housing status. Participants will be recruited in the Raleigh-Durham-Cary combined statistical area (CSA) area of North Carolina. Qualified subjects will complete a dietary questionnaire and come to the EPA Human Studies Facility for 3 sessions. The following endpoints will be taken from subjects: blood pressure, heart rate variability (HRV), venous blood, retinal imaging, and spirometry. Blood collected will be assessed for markers of inflammation, oxidative stress, vasoconstriction, coagulation, as well as nutritional status. Air pollution exposure will be assessed for the 24-hour and weeklong period of each visit using area-specific air quality data, provided by stationary air monitors. In addition, participants will be provided with silicone wrist bands to wear for three weeklong intervals during the duration of their study. Silicone wrist bands have been shown to sorb a wide range of volatile and semi-volatile compounds and will serve as a passive personal exposure monitor to air. The investigators hypothesize that residence in a neighborhood with high social vulnerability will increase both personal exposure to air pollution and the associated health effects of air pollution exposure. The investigators further hypothesize that nutrition, specifically components in nutrition demonstrated to be anti-inflammatory, will modulate this relationship and reduce cardiopulmonary outcomes associated with exposure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-70 years old males and females.
* Residing in Zip Code Tabulation Area in Raleigh-Durham great triangle area representing high or low social vulnerability index (SVI).
* Continuous residence at the same address during previous one year.

Exclusion Criteria:

* Individuals with a diagnosis of COVID-19 and have persistent symptoms due to that infection (e.g., shortness of breath) or symptoms consistent with "long COVID".
* Individuals not "up to date" on their vaccinations for COVID-19. [which means a person who has received all recommended COVID-19 vaccines, including any booster dose(s) when eligible].
* Individuals who have difficulty to come to the HSF medical station on a weekday for data collection without assistance.
* Individuals have a history of heart arrhythmia, a pacemaker user, been diagnosed with arrhythmia and prescribed a medication to treat arrhythmia.
* Individuals have uncontrolled hypertension (>180 systolic, >110 diastolic)
* Individuals who are currently smoking (including vaping, hookah, e-cigarettes, including marijuana, CBD, and/or THC products) or have a smoking history within 1 year of study (defined as more than 1 pk/yr in the past year) or have a greater than/equal to a 5-pack year smoking history.
* Individuals living with a smoker who smokes inside the house.
* Individuals who are regularly exposed to high levels of vapors, dust, gases, smoke, or fumes.
* Individuals who do not understand or speak English.
* Individuals who are taking β-blocker medications.
* Individuals who are on specific extreme diets, such as liquid diet, weight loss diet, or single diet.
* Individuals who are unwilling or unable to maintain their current dietary and medication pattern for the whole study.
* Individuals with bleeding or clotting disorders.
* Individuals who have skin allergy to tape or electrodes.
* Individuals who are pregnant or attempting to become pregnant.
* Individuals currently on dialysis
* Individuals who have unspecified illnesses, which in the judgment of the investigators might increase the risk associated with clinical procedures will be a basis for exclusion.

Temporary Exclusion Criteria :

* Individuals who have had recent (within 6 months) abdominal and/or eye surgery, or been diagnosed with any type of hernia, as well as any other contraindications for raised intra-abdominal pressure.
* Individuals who have prolonged chest pain at rest (severe uncompensated angina pectoris) or inability to carry out any physical activity without chest discomfort.
* Individuals who have difficulty breathing when at rest or performing activities at daily living.
* Individuals who are having an acute respiratory illness within two weeks prior to any of the study visits.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population represents individuals living in neighborhoods ranked either at the top or bottom of the Social Vulnerability Index, a measure of community vulnerability.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability - SDNN | Through study completion, an average of 1-2 years
  Time-domain measurement: standard deviation of the normal-to-normal (SDNN) in milliseconds
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure
Heart Rate Variability - rMSSD | Through study completion, an average of 1-2 years
  Time-domain measurement: root-mean squared of successive differences (rMSSD) in milliseconds
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure
Heart Rate Variability - LF absolute power | Through study completion, an average of 1-2 years
  Frequency-domain measurement: Low frequency power (LF, 0.04-0.15 Hz) in ms squared divided by cycles per second (ms2/Hz).
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure
Heart Rate Variability - VLF absolute power | Through study completion, an average of 1-2 years
  Frequency-domain measurement: Very Low frequency power (VLF, 0.0033-0.04 Hz) in ms squared divided by cycles per second (ms2/Hz).
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure
Heart Rate Variability - HF absolute power | Through study completion, an average of 1-2 years
  Frequency-domain measurement: High frequency power (HF, 0.15-0.40 Hz) in ms squared divided by cycles per second (ms2/Hz).
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure
Heart Rate Variability - LF/HF power | Through study completion, an average of 1-2 years
  Frequency-domain measurement: ratio of LF power divided by HF power, expressed as ratio
  This outcome is measured repeatedly to assess change in HRV associated with change in ambient air pollution exposure

SECONDARY OUTCOMES:
Pulmonary Function - FVC | Through study completion, an average of 1-2 years
  Forced vital capacity (FVC) measured in Liters (L) measured via Sensor Medic Vmax pulmonary function system (dry rolling seal spirometer).
  This outcome is measured repeatedly to assess change in lung function associated with change in ambient air pollution exposure
Pulmonary Function - FEV1 | Through study completion, an average of 1-2 years
  Forced Expiratory Volume in 1 second (FEV1) measured in Liters (L) measured via Sensor Medic Vmax pulmonary function system (dry rolling seal spirometer).
  This outcome is measured repeatedly to assess change in lung function associated with change in ambient air pollution exposure
Pulmonary Function - FEV1/FVC | Through study completion, an average of 1-2 years
  the ratio of Forced Expiratory Volume in 1 second (FEV1) measured in Liters (L) divided by Forced Vital Capacity (FVC) measured in Liters (L) measured via Sensor Medic Vmax pulmonary function system (dry rolling seal spirometer). Expressed as a percentage
  This outcome is measured repeatedly to assess change in lung function associated with change in ambient air pollution exposure
Peripheral Venous Blood - Total Cholesterol | Through study completion, an average of 1-2 years
  Total cholesterol measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in blood lipids associated with change in ambient air pollution exposure
Peripheral Venous Blood - HDL | Through study completion, an average of 1-2 years
  High density lipoproteins measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in blood lipids associated with change in ambient air pollution exposure
Peripheral Venous Blood - LDL | Through study completion, an average of 1-2 years
  Low density lipoproteins measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in blood lipids associated with change in ambient air pollution exposure
Peripheral Venous Blood - VLDL | Through study completion, an average of 1-2 years
  Very Low density lipoproteins measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in blood lipids associated with change in ambient air pollution exposure
Peripheral Venous Blood - Triglycerides | Through study completion, an average of 1-2 years
  Triglycerides measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in blood lipids associated with change in ambient air pollution exposure
Peripheral Venous Blood - CRP | Through study completion, an average of 1-2 years
  C Reactive Protein measured in plasma in milligrams per deciliter (mg/dL)
  This outcome is measured repeatedly to assess change in inflammatory markers associated with change in ambient air pollution exposure
Peripheral Venous Blood - IL1B | Through study completion, an average of 1-2 years
  Cytokine IL1B measured in plasma in picograms per milliliter (pg/mL)
  This outcome is measured repeatedly to assess change in inflammatory markers associated with change in ambient air pollution exposure
Peripheral Venous Blood - IL6 | Through study completion, an average of 1-2 years
  Cytokine IL6 measured in plasma in picograms per milliliter (pg/mL)
  This outcome is measured repeatedly to assess change in inflammatory markers associated with change in ambient air pollution exposure
Peripheral Venous Blood - IL8 | Through study completion, an average of 1-2 years
  Cytokine IL8 measured in plasma in picograms per milliliter (pg/mL)
  This outcome is measured repeatedly to assess change in inflammatory markers associated with change in ambient air pollution exposure
Peripheral Venous Blood - TNFa | Through study completion, an average of 1-2 years
  Cytokine TNFa measured in plasma in picograms per milliliter (pg/mL)
  This outcome is measured repeatedly to assess change in inflammatory markers associated with change in ambient air pollution exposure
Retinal Vasculature - CRAE | Through study completion, an average of 1-2 years
  Retinal images taken via non-mydriatic fundus camera are analyzed for central retinal artery equivalent (CRAE) measured in micrometer (um)
  This outcome is measured repeatedly to assess change in retinal vasculature associated with change in ambient air pollution exposure
Retinal Vasculature - CRVE | Through study completion, an average of 1-2 years
  Retinal images taken via non-mydriatic fundus camera are analyzed for central retinal venous equivalent (CRAE) measured in micrometer (um)
  This outcome is measured repeatedly to assess change in retinal vasculature associated with change in ambient air pollution exposure
Retinal Vasculature - AVR | Through study completion, an average of 1-2 years
  Retinal images taken via non-mydriatic fundus camera are analyzed for arteriole to venule ratio (AVR), which is central retinal venous equivalent (CRAE) measured in micrometer (um) divided by central retinal artery equivalent (CRAE). Expressed as a ratio T wave complexity

OTHER OUTCOMES:
Concentration of Air Toxics via Silicone Wrist Band | Through study completion, an average of 1-2 years
  Measurement of SVOCs sorbed to silicone wrist bands

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States